CLINICAL TRIAL: NCT05961904
Title: Impact of Breast Milk on Cortical Pain Response in Newborns During the Heel Prick Procedure: A Randomized Controlled Trial
Brief Title: Impact of Breast Milk on Cortical Pain Response in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ozgul Bulut, Principal Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Ozgul2
Record Dates: First submitted 2023-07-05; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pain Management
Keywords: Analgesia; breastmilk; cortical pain response; heal prick procedure; Near-infrared spectroscopy
MeSH Terms: conditions — Agnosia | interventions — Milk, Human

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Study group with receive orally breast milk
  Interventions: Other: Breastmilk
- Control group (No Intervention): no intervention

INTERVENTIONS:
Other: Breastmilk — Study group with receive orally 2 ml breast milk before the heel prick.
  Other Names: Human milk
  Arms: Study group

SUMMARY:
Background:Newborns are exposed to painful procedures for many different reasons in the first days of their life. If pain is not relieved effectively in these newborns, neurodevelopmental and behavioral problems may occur in the short- and long-term.

Objective:This study is aimed to investigate the effects of breast milk on cortical pain response and behavioral response in newborns during heel-prick procedure.

Design: A prospective, randomized controlled trial was conducted on newborns born in a university hospital. Healthy-term newborns, undergoing heel blood sampling for newborn screening, were enrolled in the study. Infants were randomly assigned to study group with receive orally 2 ml breast milk (n=45) or a control group with no intervention (n=45) before the heel prick. A near-infrared spectroscopy device was used to monitor regional cerebral oxygen saturation (rScO2), while neonatal pain expression was assessed by Neonatal Pain, Agitation, and Sedation Scale (N-PASS). The rScO2 measure was the primary outcome, while the N-PASS score, heart rate, SaO2, and crying time were the secondary outcomes.

DETAILED DESCRIPTION:
During the first few days of life, newborns are exposed to painful and stressful procedures.1, 2 One of these is the metabolic disease screening test using the heel-prick procedures.3, 4 Newborn screening is crucial to detect several congenital genetic and metabolic disorders at an early stage for the earliest possible recognition and management of affected newborns and to prevent morbidity, mortality, and disabilities associated with inherited metabolic disorders5. Pain induced by these procedures is ineffectively prevented or inadequately treated1. Consequently, this may have short- and long-term negative effects on the pain response and neurodevelopmental outcomes.6, 7, 8 Thus, effectively identifying, assessing, and managing neonatal pain are crucial to minimizing its impact on the intermediate- and long-term outcomes in newborns.2, 9 Near-infrared spectroscopy (NIRS) is a noninvasive technique widely used in neonatal pain research to measure functional activation of the cortex.20, 21, 22, 23 NIRS has revealed that blood sampling can activate the neonatal somatosensory20, 21, motor24, and prefrontal22 areas starting at the 25th week of postmenstrual age. Pain increases oxygen consumption with changes occurring in the primary somatosensory cortex on the brain surface.25, 26 Additionally, the relationship between the total Premature Infant Pain Profile (PIPP)27 score and hemodynamic response has been evaluated.

Among the analgesics studied for neonatal pain, breast milk is a natural substance beneficial and nutritious for infants.32 Whether breast milk administration alters cortical brain activation in neonates is presently unclear. Therefore, we conducted a trial to assess whether breast milk can relieve cortical pain during a painful metabolic disease screening procedure.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria selected neonates born after 37 weeks of gestation, postnatal age more than 24 hours (h), absence of congenital malformations, ongoing intubation, and mechanical ventilation, who had not received analgesic, anesthetic, or sedative drugs.

Exclusion Criteria:

* Neonates born before 37 weeks of gestation

Ages: 2 Days to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
The rScO2 measure was the primary outcome. | 2 months
  A near-infrared spectroscopy device was used to monitor regional cerebral oxygen saturation (rScO2). Pain increases oxygen consumption with changes occurring in the rScO2 measure.

SECONDARY OUTCOMES:
The Neonatal Pain, Agitation, and Sedation scale | 2 months
  The mean of the Neonatal Pain, Agitation, and Sedation score (A score >+3 indicates pain)

CONTACTS AND LOCATIONS:
Overall Officials: Ozgul Bulut, Principal Investigator — Istanbul Medeniyet University Goztepe Prof. Dr. Suleyman Yalcın City Hospital
Locations (1):
- Istanbul Medeniyet University Goztepe Prof. Dr. Suleyman Yalcın City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bulut O, Topaloglu SC, Bulut N, Hocaoglu M, Arslanoglu S. Impact of breast milk on cortical pain response in newborns during the heel prick procedure: a randomized controlled trial. J Perinatol. 2024 Nov;44(11):1675-1681. doi: 10.1038/s41372-024-02081-4. Epub 2024 Aug 12. PMID 39134667